CLINICAL TRIAL: NCT01305434
Title: Randomized Double Blind Cross Over Trial to Examine the Effect of Mulberry Leaf Extract on Post Prandial Glucose in Type 2 Diabetics
Brief Title: Mulberry Leaf Extract and Blood Glucose Control in Diabetics
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Craig, Nancy, M.D. (Individual)
Responsible Party: Principal Investigator, Nancy Craig, Dr. Nancy Craig, Craig, Nancy, M.D.
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: MLE-DM2
Record Dates: First submitted 2011-02-24; First posted 2011-02-28 (Estimated); Last update posted 2015-02-04 (Estimated); Status verified 2015-02

CONDITIONS: Diabetes Mellitus Type 2
Keywords: diabetes mellitus type 2; mulberry leaf extract; post prandial blood glucose
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo then mulberry leaf (Other): These patients receive placebo for two weeks, then 1 week washout, then two weeks of mulberry leaf extract.
  Interventions: Dietary Supplement: Mulberry leaf extract effect on post prandial blood glucose
- Mulberry leaf then placebo (Other): These patients receive mulberry leaf extract for two weeks, then 1 week washout, then two weeks of placebo.
  Interventions: Dietary Supplement: Mulberry leaf extract effect on post prandial blood glucose

INTERVENTIONS:
Dietary Supplement: Mulberry leaf extract effect on post prandial blood glucose — Mulberry leaf extract (400 mg, Mulberry Zuccarin, New Nordic) or placebo will be administered with meals to type 2 diabetics. Half the patients will receive mulberry leaf extract for the first two weeks and half will receive placebo. Following a one week wash out period, the interventions will be reversed for another 2 weeks, followed by a final wash out period. Subjects will keep diaries of food, exercise, daily fasting glucose, and at least one 2 hour pc glucose per day for the 6 weeks of the trial.
  Baseline renal function blood work and urine, liver function blood work, hemoglobin A1C, weight, and blood pressure will be done. These will be repeated at the end of each subject's 6 weeks in the trial. In addition, blood pressure will be checked with the distribution of the each 2 week batch of medications.
  Other Names: Mulberry Zuccarin, 400 mg tablets. New Nordic (Sweden)

SUMMARY:
Mulberry leaf teas or extracts are used as a natural remedy for diabetes in some countries. Animal studies have shown some effect of mulberry leaf extract on blood glucose. The purpose of this trial is to assess the effect of mulberry leaf extract on type 2 diabetics, by measuring blood glucose two hours after eating a meal and taking a capsule containing either mulberry leaf extract or a placebo.

DETAILED DESCRIPTION:
Patients will participate in a double blind randomized cross over trial for 6 weeks. Four 2 weeks, half of the type 2 diabetic patients will receive mulberry leaf capsules three times per day with meals (made from Mulberry Zuccarin tablets - New Nordic, 400 mg of mulberry leaf extract per tablet) and half will receive placebo capsules. Following a one week wash out period, the treatments administered to each group will be reversed for the next 2 weeks, and data will continue to be gathered for a final wash out week. Patients will keep a diary of food, exercise, and fasting glucose each morning as well as at least one 2 hour pc glucose each day. Weight, hemoglobin A1C, liver function tests, and renal function tests will be done at baseline and at the end of the 6 weeks. As well, blood pressure will be monitored when the 2 weekly batches of medication are distributed, and at the end of the 6 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Type 2 diabetes
* baseline hemoglobin A1C greater than or equal to 7.5 or fasting glucose greater than 7 (SI units)

Exclusion Criteria:

* on insulin
* history of hepatic or renal disease
* pregnant or nursing women

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-09; Primary Completion 2014-10 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
change in 2 hour post prandial blood glucose | 6 weeks
  Success would be a change in pc glucose of -1.5 units (SI) greater than 70% of the time or in more than 70% of subject, and no increased incidence of hypoglycemia with the intervention

SECONDARY OUTCOMES:
number of subjects with adverse changes in creatinine, AST, ALT, and blood pressure due to intervention | 6 weeks
  Because mulberry leaf tea has been shown to contain cadmium which can have renal or hepatotoxic effects, renal function, liver function, and blood pressure will be monitored.

CONTACTS AND LOCATIONS:
Overall Officials: Nancy V Craig, MDCM, Principal Investigator; William R Craig, MD CM, Study Director — University of Alberta
Locations (1):
- Hope Medical Clinic, Edmonton, Alberta, Canada

REFERENCES:
- [Background] Miyahara C, Miyazawa M, Satoh S, Sakai A, Mizusaki S. Inhibitory effects of mulberry leaf extract on postprandial hyperglycemia in normal rats. J Nutr Sci Vitaminol (Tokyo). 2004 Jun;50(3):161-4. doi: 10.3177/jnsv.50.161. PMID 15386927
- [Background] Park JM, Bong HY, Jeong HI, Kim YK, Kim JY, Kwon O. Postprandial hypoglycemic effect of mulberry leaf in Goto-Kakizaki rats and counterpart control Wistar rats. Nutr Res Pract. 2009 Winter;3(4):272-8. doi: 10.4162/nrp.2009.3.4.272. Epub 2009 Dec 31. PMID 20098579
- [Background] Andallu B, Varadacharyulu NCh. Antioxidant role of mulberry (Morus indica L. cv. Anantha) leaves in streptozotocin-diabetic rats. Clin Chim Acta. 2003 Dec;338(1-2):3-10. doi: 10.1016/s0009-8981(03)00322-x. PMID 14637259
- [Background] Park MY, Lee KS, Sung MK. Effects of dietary mulberry, Korean red ginseng, and banaba on glucose homeostasis in relation to PPAR-alpha, PPAR-gamma, and LPL mRNA expressions. Life Sci. 2005 Nov 12;77(26):3344-54. doi: 10.1016/j.lfs.2005.05.043. Epub 2005 Jun 23. PMID 15979095
- [Background] Naowaboot J, Pannangpetch P, Kukongviriyapan V, Kongyingyoes B, Kukongviriyapan U. Antihyperglycemic, antioxidant and antiglycation activities of mulberry leaf extract in streptozotocin-induced chronic diabetic rats. Plant Foods Hum Nutr. 2009 Jun;64(2):116-21. doi: 10.1007/s11130-009-0112-5. PMID 19434497
- [Background] Oku T, Yamada M, Nakamura M, Sadamori N, Nakamura S. Inhibitory effects of extractives from leaves of Morus alba on human and rat small intestinal disaccharidase activity. Br J Nutr. 2006 May;95(5):933-8. doi: 10.1079/bjn20061746. PMID 16611383
- [Background] Hansawasdi C, Kawabata J. Alpha-glucosidase inhibitory effect of mulberry (Morus alba) leaves on Caco-2. Fitoterapia. 2006 Dec;77(7-8):568-73. doi: 10.1016/j.fitote.2006.09.003. Epub 2006 Sep 22. PMID 17071014
- [Background] Zhong L, Furne JK, Levitt MD. An extract of black, green, and mulberry teas causes malabsorption of carbohydrate but not of triacylglycerol in healthy volunteers. Am J Clin Nutr. 2006 Sep;84(3):551-5. doi: 10.1093/ajcn/84.3.551. PMID 16960168
- [Background] Mudra M, Ercan-Fang N, Zhong L, Furne J, Levitt M. Influence of mulberry leaf extract on the blood glucose and breath hydrogen response to ingestion of 75 g sucrose by type 2 diabetic and control subjects. Diabetes Care. 2007 May;30(5):1272-4. doi: 10.2337/dc06-2120. Epub 2007 Feb 15. No abstract available. PMID 17303787
- [Background] Andallu B, Suryakantham V, Lakshmi Srikanthi B, Reddy GK. Effect of mulberry (Morus indica L.) therapy on plasma and erythrocyte membrane lipids in patients with type 2 diabetes. Clin Chim Acta. 2001 Dec;314(1-2):47-53. doi: 10.1016/s0009-8981(01)00632-5. PMID 11718678
- [Background] Nookabkaew S, Rangkadilok N, Satayavivad J. Determination of trace elements in herbal tea products and their infusions consumed in Thailand. J Agric Food Chem. 2006 Sep 6;54(18):6939-44. doi: 10.1021/jf060571w. PMID 16939361
- See also: Another trial looking at a similar question (completed but not published at the time of this protocol) — http://www.clinicaltrials.gov/ct2/show/NCT00795704?term=mulberry+leaf+extract&rank=1